CLINICAL TRIAL: NCT01400919
Title: Protege® EverFlex™ and GPS™ Self-Expanding Iliac Study (DURABILITY™ Iliac)
Brief Title: DURABILITY™ Iliac Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-5684
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Arterial Disease; Claudication
Keywords: Peripheral arterial disease; claudication; stent; EverFlex; GPS; Iliac Artery
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

ARMS (1):
- Protégé™ EverFlex™ and GPS™ Self-Expanding Stent Systems (Experimental): The objective of the study is to confirm the safety and effectiveness of the Protégé EverFlex and Protégé GPS Self-Expanding Stent Systems in the treatment of stenotic, restenotic or occluded lesions in the common and external iliac artery.
  Interventions: Device: Protégé® EverFlex™ Self-Expanding Stent System, and Protégé® GPS™ Self-Expanding Stent System.

INTERVENTIONS:
Device: Protégé® EverFlex™ Self-Expanding Stent System, and Protégé® GPS™ Self-Expanding Stent System. — Implantation of one or more study devices in the common and/or external iliac artery.

SUMMARY:
The DURABILITY Iliac study is a prospective, multi-center, non-randomized study confirming the safety and effectiveness of stenting using the Protégé® EverFlex™ and Protégé® GPS™ Self-Expanding Stent Systems for the treatment of atherosclerotic lesions in the common and/or external iliac arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient has claudication as defined by a Rutherford Clinical Category Score of 2, 3 or 4.
* Evidence of ≥ 50% stenosis, restenosis or occlusion of target lesion(s) located in the common iliac artery and/or external iliac artery.
* Willing to comply with all follow-up evaluations at the specified times.
* Provides written informed consent prior to enrollment in the study.

Exclusion Criteria:

* Previous implantation of stent(s) in the target vessel.
* Received endovascular treatment of the target lesion within six months prior to the index procedure.
* Known hypersensitivity to contrast material that cannot be adequately pretreated.
* Known hypersensitivity to nickel-titanium.
* Life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Faries, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; John H. Rundback, M.D., Principal Investigator — Holy Name Medical Center
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protégé™ EverFlex™ and GPS™ Self-Expanding Stent Systems
Started | 75
Completed | 67
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Missed visit | 2

BASELINE CHARACTERISTICS:
Arm/Group | Protégé™ EverFlex™ and GPS™ Self-Expanding Stent Systems
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event Rate
Time Frame: 9 months
Measure: Number; unit: percentage of participants
Arm/Group | Protégé™ EverFlex™ and GPS™ Self-Expanding Stent Systems
Number analyzed (Participants) | 75
percentage of participants | 1.3

ADVERSE EVENTS:
Time Frame: All events that occured within 9 months
Arm/Group | Protégé™ EverFlex™ and GPS™ Self-Expanding Stent Systems
Serious Adverse Events (participants affected / at risk) | 29/75
Other Adverse Events (participants affected / at risk) | 44/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protégé™ EverFlex™ and GPS™ Self-Expanding Stent Systems (N=75)
Cardiac disorders (Cardiac disorders) | 6 (9)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2)
General disorders and administration site conditions (General disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 7 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Nervous system disorders (Nervous system disorders) | 3 (3)
Vascular disorders (Vascular disorders) | 12 (18)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protégé™ EverFlex™ and GPS™ Self-Expanding Stent Systems (N=75)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 13 (18)
General disorders and administration site conditions (General disorders) | 14 (15)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 (15)
Vascular disorders (Vascular disorders) | 8 (8)
espiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (5)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results without permission of the sponsor.

Trial is still ongoing